CLINICAL TRIAL: NCT01687101
Title: A Study to Evaluate the Efficacy and Tolerability of STOPAIN in the Treatment of a Single Migraine Attack
Brief Title: STOPAIN in the Treatment of a Single Migraine Attack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDS/STPAIN/01
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Migraine; Headache
Keywords: acute migraine; acute migraine treatment; topical treatment
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Menthol; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STOPAIN topical gel (Experimental): STOPAIN gel which is topical menthol 6% gel applied as 2 to 4 pumps of gel applied behind the ears and to the occipital region of the neck in one or two applications within 2 hours of the onset of the migraine.
  Interventions: Drug: STOPAIN topical gel

INTERVENTIONS:
Drug: STOPAIN topical gel — STOPAIN topical gel is topical menthol 6% gel applied as 2 to 4 pumps of gel applied behind the ears and to the occipital region of the neck in one or two applications within 2 hours of the onset of the migraine.
  Other Names: Topical menthol 6% gel

SUMMARY:
This is an open label pilot study of 25 subjects with a diagnosis of episodic migraine with or without aura. STOPAIN is an over-the-counter product that is used for the temporary relief of minor aches and pains of muscles and joints associated with simple backache, arthritis, strains, bruises and sprains. We plan to have subjects apply the product during a single migraine attack to see if it will alleviate the headache pain and associated symptoms.

DETAILED DESCRIPTION:
This is an open label, 2 visit, pilot study of 25 subjects with a diagnosis of episodic migraine with or without aura according to the International Classification of Headache Disorders (2nd Edition-2004).

Subjects will be screened at Visit 1 after being properly consented for participation in the study. Screening procedures will include assessment of the medical history, headache history, current medications, vital signs, height and weight measurements and a urine pregnancy test for women of childbearing potential. Investigators will determine the eligibility of study subjects. Subjects will be instructed on how and when to apply the topical gel to treat a migraine attack. In addition, subjects will be instructed how to complete the take home diary. The study medication will be used at home to treat a single migraine attack.

At the time of at-home treatment the subject will apply the study medication. The gel will be applied to the area below and abutting the back base of the skull to base of neck and span from behind and between both ears. The quantity shall be two pumps from the metered dosing bottle. The best way to apply is to pump once onto the fingertips and apply the gel to one-half of the application area and pump again onto the fingertips and apply the gel to the other half of the application area. Massage in for 5 to 10 seconds to make sure there is reasonably uniform coverage. (Do not cover with cloth or bandage or lie down on a pillow until the gel has completely dried - about 10 minutes or so.) Do not get any of the gel into the eyes or onto mucus membranes. The gel is not toxic but will cause a burning sensation to eyes or mucus membranes. Wash hands with soap and warm water after application. The gel will give rise to a cooling sensation and to it may feel like a mild to moderate stinging or burning sensation. That is normal. Anything more than a mild to moderate stinging or burning sensation is not expected and should be noted in diary. If there has been no reduction in symptoms after 30 minutes repeat the application. If there is no relief after 2 hours the subject may use other rescue medication.

Completed subject diaries will provide data on headache severity and the presence or absence of nausea, vomiting, photophobia and phonophobia. Time of resolution of both the headache and accompanying symptoms will be collected. The subjects will record migraine pain severity and the presence or absence of associated symptoms at 30, 60, 90 minutes and 2, 4, and 24 hours after the administration of study drug.

Subjects will be asked to treat a single migraine attack within 8 weeks of Visit 1. After treating the attack and completing the diary, they will be asked to return to Jefferson Headache Center for a final visit (Visit 2) or to return the diary and other study supplies by mail. Shipping materials will be provided to each participant.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 and 65, inclusive
* Subjects diagnosed with episodic migraine, with or without aura according to IHS criteria for at least one year prior to screening
* Subjects who experience between 1 and 10 migraine attacks (inclusive) per month (during the previous 6 months) with no more than 15 days of headache per month.
* Subject is using or agrees to use for the duration of participation a medically acceptable form of contraception (as determined by investigator), if female of child-bearing potential
* Subjects who are able to understand and comply with all study procedures.
* Subject provides written informed consent prior to any screening procedures being conducted

Exclusion Criteria:

* Pregnant and/or lactating women
* Subjects who, in the investigator's opinion, have a history or have evidence of a medical or psychiatric condition that would expose them to an increased risk of a significant adverse event or would interfere with the assessments of efficacy and tolerability during this trial
* Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit
* Subjects who currently have or have had a history of basilar or hemiplegic migraine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Silberstein, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | STOPAIN Topical Gel
Started | 32
Completed | 25
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | STOPAIN Topical Gel
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of STOPAIN in the Acute Treatment of Migraine
Description: To evaluate the efficacy of STOPAIN in the acute treatment of migraine as measured by Pain Freedom (headache pain intensity level equal to "no pain") at 2 hours post dose using a four point numeric rating scale (0=no pain, 1= mild pain, 2=moderate pain, 3=severe pain).
Time Frame: 2 hours after the time of gel application
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | STOPAIN Topical Gel
Number analyzed (Participants) | 25
units on a scale | 1.92 [0 to 3]

ADVERSE EVENTS:
Time Frame: 24 hours after application of topical gel.
Arm/Group | STOPAIN Topical Gel
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 2/32
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STOPAIN Topical Gel (N=32)
Stinging (Skin and subcutaneous tissue disorders) | 1 (1) — Stinging at application site resolved without treatment. Duration of 15 minutes.
Burning sensation. (Skin and subcutaneous tissue disorders) | 1 (1) — Burning sensation on both hands after applying gel. Duration 20 minutes; severity was mild. Resoved without treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes